CLINICAL TRIAL: NCT00002425
Title: A Multicenter, Open-Label Study of the Safety and Activity of Saquinavir Soft Gelatin Capsule Formulation (Saquinavir SGC) in Combination With Other Antiretroviral Drugs
Brief Title: The Safety and Effectiveness of Saquinavir Soft Gelatin Capsules Combined With Other Anti-HIV Drugs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 229E; NV15182B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-12

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Saquinavir; HIV Protease Inhibitors; Dosage Forms; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Saquinavir

INTERVENTIONS:
Drug: Saquinavir

SUMMARY:
To evaluate the safety and antiretroviral activity of saquinavir soft gelatin capsule formulation (SQV-SGC) in combination with other antiretroviral drugs.

DETAILED DESCRIPTION:
All patients receive SQV as monotherapy or in combination with other antiretroviral drugs chosen by the investigator and patient. (This study provides only SQV.) Patients may not choose another protease inhibitor (PI) as part of their combination therapy; furthermore, patients taking PIs other than SQV must undergo a 5-day washout period before study-drug administration. Patients are monitored for adverse events and changes in routine laboratory tests, plasma viral load, and CD4+ T cell levels. Outcomes are analyzed by stratifying patients according to CD4+ T cell levels and prior history with protease inhibitors.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

Antiretroviral treatments other than PIs.

Patients must have:

* HIV infection.
* No prior experience with PIs. (Note:
* At least 75 percent of patients must be naive to PIs.)

Exclusion Criteria

Concurrent Medication:

Excluded:

PIs other than SQV.

Prior Medication:

Excluded:

Any PIs (see note in General Criteria--Inclusion).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400

CONTACTS AND LOCATIONS:
Locations (1):
- Consumer Contact, Nutley, New Jersey, United States